CLINICAL TRIAL: NCT03485924
Title: Endoscopic Ultrasound With Fine Needle Biopsy Versus Fine Needle Aspiration With On-Site Cytopathology in the Evaluation of Solid Pancreatic Masses: Randomized Single Blinded Clinical Trial
Brief Title: EUS FNB Versus FNA With On-Site Cytopathology in Solid Pancreatic Masses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is not relevant anymore.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB00148609
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Fine Needle Aspiration; Pancreatic Mass
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EUS-FNA with ROSE (Active Comparator): EUS/FNA with ROSE will be performed using standard techniques via 22-g FNA needle (Cook Medical EchoTip Ultra or Boston Scientific Expect or Medtronic Beacon). Lesions will be identified using EUS and punctured with the FNA needle (10-15 back and forth movements per needle pass, fanning as appropriate). After the lesion is punctured, the stylet will be removed and 10cc suction will be applied. FNA specimens will be processed for ROSE using standard techniques with bedside smear slide evaluation and liquid-based cytology and cell-block preparation.
  Interventions: Diagnostic Test: EUS-FNA with ROSE
- EUS-FNB without ROSE (Active Comparator): EUS/FNB without ROSE will be performed using similar techniques for tissue acquisition as FNA using 22-g FNB needle (Medtronic SharkCore or Boston Scientific Acquire). Lesions will be identified using EUS and punctured with the 22-g FNB needle (10-15 back and forth movements per needle pass, fanning as appropriate). After the lesion is punctured, the stylet will be removed and 10cc suction will be applied. FNB samples will be placed directly into formalin containers and sent to be processed by surgical pathology.
  Interventions: Diagnostic Test: EUS-FNB without ROSE

INTERVENTIONS:
Diagnostic Test: EUS-FNA with ROSE — EUS-FNA with ROSE vs EUS-FNB without ROSE
  Arms: EUS-FNA with ROSE
Diagnostic Test: EUS-FNB without ROSE — EUS-FNA with ROSE vs EUS-FNB without ROSE
  Arms: EUS-FNB without ROSE

SUMMARY:
The objective of this paired cohort study is to evaluate the diagnostic accuracy of Endoscopic Ultrasound-fine needle aspiration (EUS-FNA) with rapid onsite evaluation (ROSE) compared to EUS-fine needle biopsy (EUS-FNB) without ROSE. If EUS-FNB without ROSE is shown to be non-inferior to the current standard of care of EUS-FNA with ROSE in pancreatic lesions, this study has the potential to make EUS-guided tissue acquisition more economical (with elimination for the need for cytopathology staff onsite) as well as provide core histological specimen without sacrificing the overall diagnostic yield.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) guided fine needle aspiration (EUS-FNA) is the primary technique for tissue acquisition for pancreatic lesions. Despite widespread adoption of the techniques, the diagnostic yield of EUS-FNA for pancreatic lesion is highly variable, with sensitivities ranging from 64-95%, specificities ranging from 75-100% and overall diagnostic accuracy ranging from 78-95%.

Despite its mainstay as the primary technique for tissue acquisition, EUS-FNA has several limitations. The standard EUS-FNA does not routinely provide core biopsy specimen with preserved tissue architecture, which is required for immunohistochemical staining and for definitive diagnosis of conditions, such as lymphoma, gastrointestinal stromal tumors, Immunoglobulin G (IgG)-4-associated lymphoplasmacytic sclerosing pancreatitis. Furthermore, the diagnostic yield of EUS-FNA is highly dependent on the availability of bedside cytotechnologist or cytopathologist for rapid onsite evaluation (ROSE), which increases the overall cost required to perform EUS-FNA.

Recently, multiple dedicated EUS fine needle biopsy (FNB) needles have been developed to obtain core specimens. Early small studies have shown promising results with these EUS-FNB needles.

The objective of this paired cohort study is to evaluate the diagnostic accuracy of EUS-FNA with ROSE compared to EUS-FNA with ROSE. Participants will be assigned to the arms. If EUS-FNB without ROSE is shown to be non-inferior to the current standard of care of EUS-FNA with ROSE in pancreatic lesions, this study has the potential to make EUS-guided tissue acquisition more economical (with elimination for the need for cytopathology staff onsite) as well as provide core histological specimen without sacrificing the overall diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age referred for EUS-guided biopsy for pancreatic mass lesions

Exclusion Criteria:

* Refusal to consent form
* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Uncooperative patients
* Pregnant women (women of childbearing age will undergo urine pregnancy testing, which is routine for all endoscopic procedures)
* Medically unstable for sedation
* Entirely cystic lesions
* Lesions inaccessible to EUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EUS-FNA With ROSE: EUS/FNA with ROSE will be performed using standard techniques via 22-g FNA needle (Cook Medical EchoTip Ultra or Boston Scientific Expect or Medtronic Beacon). Lesions will be identified using EUS and punctured with the FNA needle (10-15 back and forth movements per needle pass, fanning as appropriate). After the lesion is punctured, the stylet will be removed and 10cc suction will be applied. FNA specimens will be processed for ROSE using standard techniques with bedside smear slide evaluation and liquid-based cytology and cell-block preparation. The first randomization assigned EUS sampling technique will be used until adequate specimen is achieved (up to 3 passes total). After 3 passes, the patient will undergo the other EUS sampling technique until adequate specimen is achieved (up to 3 passes total).
  EUS-FNA with ROSE: EUS-FNA with ROSE vs EUS-FNB without ROSE
- EUS-FNB Without ROSE: EUS/FNB without ROSE will be performed using similar techniques for tissue acquisition as FNA using 22-g FNB needle (Medtronic SharkCore or Boston Scientific Acquire). Lesions will be identified using EUS and punctured with the 22-g FNB needle (10-15 back and forth movements per needle pass, fanning as appropriate). After the lesion is punctured, the stylet will be removed and 10cc suction will be applied. FNB samples will be placed directly into formalin containers and sent to be processed by surgical pathology. The first randomization assigned EUS sampling technique will be used until adequate specimen is achieved (up to 3 passes total). After 3 passes, the patient will undergo the other EUS sampling technique until adequate specimen is achieved (up to 3 passes total).
  EUS-FNB without ROSE: EUS-FNA with ROSE vs EUS-FNB without ROSE
Period: Overall Study
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
Started | 23 | 17
Completed | 23 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.39 (9.95) | 69.94 (8.41) | 67.32 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 18 | 12 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: The Diagnostic Accuracy of Fine-needle Biopsy (FNB) Sampling Without Rapid Onsite Evaluation (ROSE) and the Fine Needle Aspiration (FNA) With ROSE in Pancreatic Mass Lesions
Description: Diagnostic accuracy will be defined as (true positive + true negative)/all participants in the arm.
Time Frame: 6 months from the initial biopsy
Measure: Number; unit: percentage of true cases
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
Number analyzed (Participants) | 23 | 17
percentage of true cases | 91.3 | 94.1

2. Secondary Outcome: Specimen Adequacy
Description: Number of Specimens with Final Histopathological Diagnosis
Time Frame: Post-procedure one week
Measure: Count of Units; unit: Samples
Units Other Than Participants: Samples
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
Number analyzed (Participants) | 23 | 17
Number analyzed (Samples) | 59 | 47
Samples | 35 | 47

3. Secondary Outcome: Number of Histology Cores Obtained
Description: Number of Samples with Visible Histology Core Biopsy
Time Frame: Post-procedure one week
Measure: Count of Units; unit: Samples
Units Other Than Participants: Samples
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
Number analyzed (Participants) | 23 | 17
Number analyzed (Samples) | 59 | 47
Samples | 3 | 46

4. Secondary Outcome: Median Number of Passes
Description: Median number of passes required for accurate diagnosis
Time Frame: 6 months from the initial biopsy
Population: Participants with accurate diagnosis
Measure: Median (Full Range); unit: passes
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
Number analyzed (Participants) | 21 | 16
passes | 2 [1 to 3] | 1 [1 to 1]

5. Secondary Outcome: Number of Technical Failures
Description: Technical failure was defined as the inability to perform the procedure, including the need to change the needle
Time Frame: After the procedure, an average of 1 hour
Measure: Count of Units; unit: Procedures
Units Other Than Participants: Procedures
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
Number analyzed (Participants) | 23 | 17
Number analyzed (Procedures) | 59 | 47
Procedures | 0 | 0

ADVERSE EVENTS:
Time Frame: pre, intra- and immediately post-procedure, an average of 1 hour
Arm/Group | EUS-FNA With ROSE | EUS-FNB Without ROSE
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/17
Other Adverse Events (participants affected / at risk) | 0/23 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT03485924/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03485924/ICF_001.pdf